CLINICAL TRIAL: NCT04139395
Title: 68Ga Citrate PET/MRI for Evaluation of Fever of Unknown Origin (FUO)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Not feasible at this time.
Sponsor: Carina Mari Aparici (Other)
Responsible Party: Sponsor-Investigator, Carina Mari Aparici, Clinical Professor, Radiology/ Nuclear Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-49104
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Fever of Unknown Origin
MeSH Terms: conditions — Fever of Unknown Origin | interventions — gallium citrate; Positron-Emission Tomography; Magnetic Resonance Imaging; Tomography, Emission-Computed, Single-Photon; Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic 68Ga-Citrate PET/MRI Imaging (Experimental): Participants will receive separate scans, first a SPECT scan following administration of the 67Ga Citrate tracer (standard of care), then a PET/MRI scan following administration of the 68Ga-Citrate tracer (investigational); some participants will also receive IV gadolinium-based contrast injection. Scans will be performed 45-60 minutes following injection of the tracer.
  Interventions: Drug: 68Ga-Citrate PET/MRI; Drug: 67Ga-Citrate SPECT; Device: Positron Emission Tomography; Device: Magnetic Resonance Imaging; Device: SPECT

INTERVENTIONS:
Drug: 68Ga-Citrate PET/MRI — Participants will be injected intravenously (IV) with 370 MBq of 68Ga Citrate. 45 -60 minutes after the radiopharmaceutical IV administration, whole body data acquisition at the PET/MRI suite will begin.
  Other Names: Gallium-68- Citrate
Drug: 67Ga-Citrate SPECT — 67Ga-Citrate will be used as the radiotracer for a regular medical care SPECT scan
  Other Names: Gallium-67- Citrate
Device: Positron Emission Tomography — Imaging with 68Ga-Citrate PET/MRI
  Other Names: PET
Device: Magnetic Resonance Imaging — Imaging with 68Ga-Citrate PET/MRI
  Other Names: MRI; Medical Imaging, Magnetic Resonance/ Nuclear Magnetic Resonance
Device: SPECT — Imaging with 67Ga-Citrate radiotracer. SPECT scan will be conducted as part of regular medical care.
  Other Names: Single Photon Emission Computed Tomography/Computed Tomography

SUMMARY:
This is a Phase III study to evaluate 68Ga Citrate PET/MRI for detection of origin of fever of unknown origin.

DETAILED DESCRIPTION:
The purpose of this research study is to evaluate a PET tracer (68Ga-Citrate) that can localize the origin of patients diagnosed with fever of unknown origin (FUO) using a PET/MRI scanner. We hope to learn if this can detect FUO better than with the present nuclear imaging standard of care (67Ga SPECT).

We propose the following aim:

• To evaluate 68Ga Citrate PET/MRI for detection of origin of fever in patients with fever of unknown origin.

Patients disgnosed with fever of unknown origin are injected intravenously (IV) with 370 MBq of 68Ga Citrate. 45-60 minutes later, a whole body PET/MRI images are obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patient is >/=18 years old at the time of the scan.
* Patient with diagnosis of FUO.
* Patient is capable of complying with study procedures.
* Patient can remain still for duration of imaging procedure.
* Able to provide written consent.

Exclusion Criteria:

* Patient is pregnant or nursing.
* Metallic implants (contraindicated for MRI).
* History of renal insufficiency (only for MRI contrast administration).
* Inability to lie still for the entire imaging time.
* Inability to complete the needed investigational and standard of care imaging examinations due to other reasons (severe claustrophobia, radiation phobia, etc.).
* Any additional medical condition, serious intercurrent illness, or other extenuating circumstance that, in the opinion of the investigator, may significantly interfere with study compliance.
* Known allergy, hypersensitivity, or intolerance to the investigational product or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-12-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Uptake detected by investigational imaging agent | Up to 12 months
  The uptake detected on 68Ga Citrate PET/MRI and conventional 67Ga Citrate SPECT will be compared. Outcome will be reported as infectious uptake detected per patient for each imaging method.

CONTACTS AND LOCATIONS:
Overall Officials: Carina Mari Aparici, MD, Principal Investigator — clinical professor
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No